CLINICAL TRIAL: NCT00433524
Title: Evaluation of Esophageal Motion by Computed Tomography (CT) During the Course of Thoracic Radiotherapy
Brief Title: Computed Tomography in Detecting Movement of the Esophagus in Patients Undergoing Radiation Therapy to the Chest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000304723; P30CA006927 (NIH); FCCC-03604
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Procedure: computed tomography

SUMMARY:
RATIONALE: Comparing results of diagnostic procedures, such as computed tomography scan (CT scan), done before and after radiation therapy to help detect movement of the esophagus may help doctors plan the best treatment.

PURPOSE: This clinical trial is using CT scan to help detect movement of the esophagus in patients undergoing radiation therapy to the chest.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the inter- and intra-fraction movement of the esophagus using CT scans in patients undergoing thoracic radiotherapy.

OUTLINE: This is a pilot study.

Patients undergo CT scans at baseline and then once weekly during their scheduled radiotherapy sessions to determine esophageal placement while in the treatment position. CT scans are performed before and after the radiotherapy session. Pretreatment and post-treatment scans are compared.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Planning to undergo definitive thoracic radiotherapy

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No concurrent palliative thoracic radiotherapy

Surgery

* Not specified

Other

* Concurrent participation in other clinical trials allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Inter- and intra-fraction movement of the esophagus as measured by CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Andre A. Konski, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States